CLINICAL TRIAL: NCT04490577
Title: Comparison of the Effects of Whole-Body Vibration Training and Pilates Exercises on Physical Fitness, Fatigue and Physical Self Perception in Healthy Women
Brief Title: Whole-Body Vibration Training and Pilates Exercises for Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ozlem Yuruk, PT, PHD, Assoc Prof, Baskent University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: KA18/268
Record Dates: First submitted 2020-07-07; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Healthy Lifestyle; Body Weight; Fatigue
Keywords: exercise; Physical fitness; Health
MeSH Terms: conditions — Body Weight; Fatigue; Motor Activity | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: The 36 healthy participants divided into three groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates training group (Experimental): In the Pilates group, the exercises were performed with "Reformer®" for eight weeks, twice in a week, one hour per day.
  Interventions: Other: Pilates exercises
- Whole-body vibration (WBV) group (Experimental): In the WBV group, the training was given "Power Plate®" for eight weeks, twice in a week, and 30 minutes in a day.
  Interventions: Other: Whole body vibration
- Control group (No Intervention): The control group did not receive any training.

INTERVENTIONS:
Other: Pilates exercises — Pilates exercises are a combined exercise procedure including strengthening and stretching. Pilates exercises are performed with different equipment for example; therabands, mats, reformer, etc.
  Arms: Pilates training group
Other: Whole body vibration — Whole-body vibration gives vibration to the body with a platform at different frequencies (Power-plate). The participant performed exercises on the platform.
  Arms: Whole-body vibration (WBV) group

SUMMARY:
This study aimed to compare the effects of whole-body vibration (WBV) training and Pilates exercises on physical fitness, fatigue, and physical self-perception in healthy women. This study was carried out on 36 healthy sedentary female subjects. Subjects were divided into three groups; Pilates training group, WBV training group, and control group. In the Pilates group, the exercises were performed with "Reformer®" for eight weeks, twice in a week, 45-min per day. In the WBV group, the training was given "Power Plate®" for eight weeks, twice in a week, and 30 minutes in a day. The control group did not receive any training.

DETAILED DESCRIPTION:
This study aimed to compare the effects of whole-body vibration (WBV) training and Pilates exercises on physical fitness, fatigue, and physical self-perception in healthy women aged between 25-45 years. The study was conducted between August 2018-January 2019 in a health and physiotherapy clinic. This study was carried out on 36 healthy sedantary female subjects.

Before starting the study, the subjects were divided into three groups in a randomized manner using "Random Online Allocation Software" (www.Graphpad.com)

1. Group 1: Pilates training group
2. Group 2: WBV training group
3. Group 3: Control group

Pilates training group: The exercises were performed with "Reformer®" for eight weeks, twice in a week, 45-min per day. Warm-up and cool-down exercises were performed before and after the training.

WBV training group: The training was given "Power Plate®" for eight weeks, twice in a week, and 30 minutes in a day. Warm-up and cool-down exercises were performed before and after the training.

Control group: The control group did not receive any training.

The body composition of the subjects was evaluated with body mass index, waist-hip ratio and bioelectrical impedance analysis; functional capacity with Shuttle Run Test; core endurance with lateral bridge test, modified Biering-Sorensen test, trunk flexion test and prone bridge test and functional core strength with sit-ups and modified push-up tests. The stability of the core muscles was also measured with a pressure biofeedback instrument. The Sit and Reach test was used to assess flexibility and the Functional Reach Test was used for balance. Fatigue was evaluated with The Fatigue Severity Scale and physical self-perception was assessed with the Physical Self Perception Profile. The subjects were evaluated pre-intervention and immediately after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals have not been exercising regularly in the last six months
* Physical activity level was between 600-3000 MET min/week (Metabolic equivalent minutes/week) according to the result of the "International Physical Activity Questionnaire"
* Bodyweight of less than 130 kg Individuals.

Exclusion Criteria:

* History of malignancy
* Pregnant individuals
* Musculoskeletal pain due to orthopedic or rheumatic diseases
* History of fractures in the past year
* Neurological disease (stroke, epilepsy, etc.)
* Chronic kidney or liver disease, cardiovascular diseases (cardiac arrhythmia, cardiac insufficiency, etc.)
* Imbalance due to peripheral vestibular disorder diagnosis (Benign paroxysmal positional vertigo, Meniere's disease, etc.)
* Individuals who not be able to tolerate vibration for more than five minutes were not included in the study

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Body Composition Change | Pre-intervention and immediately after the intervention
  The body composition of the subjects was evaluated with bioelectrical impedance analysis (Tanita BC 601,Tanita Corp., Maeno-Cho, Tokyo, Japan). Body fat proportion was recorded as a percentage.

SECONDARY OUTCOMES:
Body Mass Index | Pre-intervention and immediately after the intervention
  The body composition of the subjects was evaluated with body mass index (BMI). The BMI is a person's weight in kilograms divided by the square of height in meters. A high BMI can be an indicator of high body fatness.
Waist-hip ratio | Pre-intervention and immediately after the intervention
  The body composition of the subjects was also evaluated with waist-hip ratio. The waist to hip ratio measurement is calculated by dividing the measurement of your waist by your hip measurement. The score recorded as centimeter.
Aerobic capacity | Pre-intervention and immediately after the intervention
  The aerobic capacity of the participants was evaluated with Shuttle-run test. Shuttle run test involve repetitive running back and forth, either over the same distance, or with changing distances. The shorter trial recorded as seconds.
Flexibility | Pre-intervention and immediately after the intervention
  The sit and reach test used for flexibility. Sit and reach test measures measures the flexibility of the lower back and hamstring muscles.The score is recorded to the nearest centimeter as the distance reached by the hand.
Balance | Pre-intervention and immediately after the intervention
  The balance was evaluated by Functional reach test. The test evaluated dynamic balance and limit of stability. This test measures the distance between the length of an outstretched arm in a maximal forward reach from a standing position,while maintaining a fixed base of support. The score recorded as centimeter. Higher scores indicate good level of balance.
Physical Self-Perception | Pre-intervention and immediately after the intervention
  Physical self-perception was assessed with Physical Self Perception Profile. The questionnaire has four subdomain subscales designed to assess perceived bodily attractiveness, sports competence, physical strength, and physical conditioning were constructed along with a general physical self-worth subscale as the basis of the Physical Self-Perception Profile.
Fatigue Severity Scale | Pre-intervention and immediately after the intervention
  The 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle. Each item consists of statements that are scored on a seven-point Likert type scale ranging from 1 ("strongly disagree") to 7 ("strongly agree"). The higher scores indicates severe fatigue.
Lateral Bridge test | Pre-intervention and immediately after the intervention
  Lateral bridge test involves static, isometric contractions of the lateral muscles on each side of the trunk that stabilize the spine. The score recorded as second. Higher scores indicate good level of endurance.
Modified Biering-Sorensen test | Pre-intervention and immediately after the intervention
  Modified Biering-Sorensen test measuring how many seconds the subject is able to keep the unsupported upper body (from the upper border of the iliac crest) horizontal, while placed prone with the buttocks and legs fixed to the couch by three wide canvas straps and the arms folded across the chest. The score recorded as second. Higher scores indicate good level of endurance.
Trunk flexion test | Pre-intervention and immediately after the intervention
  Trunk flexion test involving a static, isometric contraction of the anterior muscles, stabilizing the spine until the individual exhibits fatigue and can no longer hold the assumed position. The score recorded as second. Higher scores indicate good level of endurance.
Prone bridge test | Pre-intervention and immediately after the intervention
  The prone bridge test measures the muscular endurance of the abdominal muscles.The score recorded as second. Higher scores indicate good level of endurance.
Sit-ups test | Pre-intervention and immediately after the intervention
  The sit-ups test is a measure the endurance of the abdominal and hip-flexor muscles. The aim of this test is to perform as many sit-ups as you can in two minutes.
Modified push-up test | Pre-intervention and immediately after the intervention
  The modified push-up test was used to measure upper body strength endurance and trunk stability. This variation, which uses a modified technique with a clap behind the back while in the 'down' position and a touch from one hand to the other in the 'up' position.The total number of correctly completed push-ups were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Yuruk, Assoc. Prof., Study Director — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)